CLINICAL TRIAL: NCT05280379
Title: Trained Immunity of Myeloid Cells and Their Progenitors in Patients With Non-medullary Thyroid Carcinoma and Colon Carcinoma
Brief Title: Trained Immunity in Thyroid Carcinoma and Colon Carcinoma
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL79885.091.21
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Cancer, Nonmedullary; Colon Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with non-medullary thyroid carcinoma: 30 patients with non-medullary thyroid carcinoma, who are going to get surgery
  Interventions: Other: no intervention will take place
- Participants with colon carcinoma: 30 participants with colon carcinoma, who are going to get surgery
  Interventions: Other: no intervention will take place

INTERVENTIONS:
Other: no intervention will take place — no intervention will take place

SUMMARY:
Tumor-related inflammation is one of the hallmarks of cancers in general. Innate immunity specifically is a common denominator which is involved in the pathogenesis of both thyroid carcinoma and colon carcinoma. To improve the patient's outcome and identify novel therapeutic targets, one needs a deeper understanding of the tumor-induced changes in the bone marrow myeloid progenitor cells. Furthermore, treatment of these cells by nanoparticles or other agents that induce a program of 'trained immunity' may be a novel way to re-educate myeloid cells and their bone marrow progenitors in thyroid carcinoma patients. Lastly, the investigators expect that this approach could be effective also in other cancers of which colon carcinoma is here proposed as an additional model.

The investigators hypothesize that by exposing myeloid cells or their progenitors to various agents that induce trained immunity (e.g. high-density-lipoprotein-methylene diphosphonate nanoparticles, recombinant and synthetic cytokines), these immune cells will undergo functional reprogramming to induce a tumor-suppressive phenotype. In the future, this could be explored as a novel immunotherapy for tumors that are refractory to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and mentally competent
* Newly diagnoses non-medullary thyroid carcinoma or colon carcinoma that is therapy naïve
* Planned to receive conventional treatment for the malignancy by surgery

Exclusion Criteria:

* Mentally incompetent
* Pregnant or breastfeeding
* Known inflammation or infectious disease or an immunosuppressive status
* Using medication interfering with the immune system
* Reduced platelets counts or other conditions associated with an increased risk of bleeding
* Severe comorbidities: other active malignancy (except for basal cell carcinoma and other in situ carcinomas)
* Previous anti-cancer treatment, such as chemotherapy, radiotherapy or surgical removal or the primary tumor
* Serious psychiatric pathology
* A self-reported alcohol consumption of >21 units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 30 participants with active colon carcinoma and 30 participants with active non-medullary thyroid carcinoma. All participants will undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Levels of pro-inflammatory cytokines en chemokines | After 7 days.
  Levels of pro-inflammatory cytokines en chemokines such as tumor necrosis factor-alfa,interleukin(IL)-1beta and IL-6 will be measured (pg/miliLiter) before and after induction of trained immunity. This will happen after 1 and after 7 days. These will be measured using ELISA.

OTHER OUTCOMES:
Age of subjects | At baseline
  Age in years of subjects
Length of subjects | At baseline
  Length in meters of subjects
Weight of subjects | Through study completion, an average of 1 year
  Weight in kilograms of subjects
Thyroid stimulating hormone | At baseline
  Levels of thyroid stimulating hormone (TSH), measured in mili unit/Liter. Only measured in the patients with thyroid carcinoma.
Carcino-embryonal antigen | At baseline
  Levels of carcino-embryonal antigen (CEA), measured in ug/Liter. Only measured in patients with colon carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No